CLINICAL TRIAL: NCT01778985
Title: Effect of Preoperative Estrogen Treatment on Connective Tissues of the Pelvic Floor
Acronym: PET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: American Urogynecologic Society Foundation Astellas Research Award (Unknown)
Responsible Party: Principal Investigator, David Rahn, MD, Assistant Professor, Dept. of Obstetrics & Gynecology, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: STU-042011-101
Record Dates: First submitted 2013-01-23; First posted 2013-01-29 (Estimated); Results first posted 2014-09-10 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-09

CONDITIONS: Pelvic Organ Prolapse; Menopause
Keywords: Pelvic organ prolapse; Menopause; Estrogen; Premarin
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Estrogens, Conjugated (USP)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Premarin (Experimental): Premarin cream 0.625mg/1gm. Applied to vagina by applicator as 1gm nightly for 2 weeks then 1gm 2 nights per week for 4-6 weeks or until day of surgery.
  Interventions: Drug: Premarin
- Placebo (Placebo Comparator): Placebo cream, applied to vagina by applicator as 1gm nightly for 2 weeks then 1gm 2 nights per week for 4-6 weeks or until day of surgery.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Premarin
  Other Names: Conjugated equine estrogen
  Arms: Premarin
Other: Placebo
  Other Names: Placebo cream
  Arms: Placebo

SUMMARY:
This is a study to determine how vaginal estrogen cream given for several weeks before pelvic reconstructive therapy will effect elastic fiber assembly in the muscularis layer of the vaginal wall. Postmenopausal women with at least Stage 2 pelvic organ prolapse will receive either estrogen vaginal cream or placebo cream 6-8 weeks prior to reconstructive surgery. At time of surgery, full thickness biopsies will be obtained from a standardized location at the top of vagina. The investigators will measure the thickness of the vaginal muscularis, elastic fiber number and morphology, and analyze if elastic fiber synthesis or degradation is affected by estrogen therapy. The results will provide important data to support a larger clinical trial to determine if preoperative and maintenance estrogen therapy alter long-term success rates of pelvic reconstructive surgery for pelvic organ prolapse.

ELIGIBILITY:
Inclusion Criteria:

* Women, still with uterus, planning total hysterectomy as part of surgical repair for pelvic organ prolapse
* Symptomatic anterior and/or apical vaginal prolapse greater than or equal to Stage 2 (i.e., bulge extends to at least 1 cm of the hymen or beyond)
* Women between 1 and 10 years after menopause. Menopause is defined as one year of amenorrhea or surgical ovariectomy.
* Age 40-70 years old
* No estrogen replacement therapy in the last 1 month
* Physically capable of daily application of vaginal cream

Exclusion Criteria:

* BMI >35
* Prior surgical repair of prolapse involving the vaginal cuff.
* Prior total hysterectomy
* Premenopausal or postmenopausal >10 years
* Prior steroid hormone replacement therapy of duration >1 month (oral or vaginal estrogen, testosterone or corticosteroids)
* History of connective tissue disease (Ehlers-Danlos, Marfan, etc)
* History of vaginal radiation
* Contraindications for estrogen replacement therapy (current, or history of, spontaneous deep vein thrombosis, stroke, coronary artery disease, breast or endometrial cancer)
* Concurrent use of steroid cream for treatment of Lichen sclerosis
* Recent history (within last month) of vaginal infection or vaginitis
* Current tobacco use

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-12; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Rahn DD, Good MM, Roshanravan SM, Shi H, Schaffer JI, Singh RJ, Word RA. Effects of preoperative local estrogen in postmenopausal women with prolapse: a randomized trial. J Clin Endocrinol Metab. 2014 Oct;99(10):3728-36. doi: 10.1210/jc.2014-1216. Epub 2014 Jun 20. PMID 24947034

RESULTS

PARTICIPANT FLOW:
Groups:
- Premarin: Premarin cream 0.625mg/1gm. Applied to vagina by applicator as 1gm nightly for 2 weeks then 1gm 2 nights per week for 4-6 weeks or until day of surgery.
  Premarin
- Placebo: Placebo cream, applied to vagina by applicator as 1gm nightly for 2 weeks then 1gm 2 nights per week for 4-6 weeks or until day of surgery.
  Placebo
Period: Overall Study
Arm/Group | Premarin | Placebo
Started | 15 | 15
Completed | 8 | 12
Not Completed | 7 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 2 | 2
Not completed — Protocol Violation | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Premarin | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (5.4) | 58.9 (5.1) | 57.2 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Hispanic White | 7 | 2 | 9
  Non-Hispanic Black | 1 | 3 | 4
  Hispanic White | 7 | 10 | 17
Parity [Median (Inter-Quartile Range); unit: deliveries] | 3 [2 to 4] | 4 [3 to 6] | 4 [3 to 6]
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 29.2 (5.4) | 31.7 (4.1) | 30.5 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Vaginal Wall Composition: Epithelium (Intention to Treat)
Description: Will assess vaginal wall histology - thicknesses of epithelium
Time Frame: Time of surgery, i.e. after 6-8 weeks of intervention
Population: Patients completing surgery with biopsy specimens available for analysis ("intention to treat")
Measure: Mean (Standard Error); unit: microns
Arm/Group | Premarin | Placebo
Number analyzed (Participants) | 12 | 12
microns | 413.9 (63.7) | 314.1 (42.6)
Statistical Analysis 1: Comparison: Premarin vs Placebo; Test type: Superiority or Other; p = 0.21, t-test, 2 sided

2. Primary Outcome: Vaginal Wall Composition: Epithelium (Per-Protocol)
Description: Will assess vaginal wall histology - thicknesses of epithelium
Time Frame: Time of surgery, i.e. after 6-8 weeks of intervention
Population: Patients completing surgery with biopsy specimens available for analysis and who were adherent to study medication ("per protocol")
Measure: Mean (Standard Error); unit: microns
Arm/Group | Premarin | Placebo
Number analyzed (Participants) | 8 | 12
microns | 550.5 (45.1) | 314.1 (42.6)
Statistical Analysis 1: Comparison: Premarin vs Placebo; Test type: Superiority or Other; p = 0.002, t-test, 2 sided

3. Primary Outcome: Vaginal Wall Composition: Muscularis (Intention to Treat)
Description: Will assess vaginal wall histology - thicknesses of muscularis
Time Frame: Time of surgery, i.e. after 6-8 weeks of intervention
Population: Patients completing surgery with biopsy specimens available for analysis ("intention to treat")
Measure: Mean (Standard Error); unit: microns
Arm/Group | Premarin | Placebo
Number analyzed (Participants) | 12 | 12
microns | 5670.4 (2154.7) | 2807.1 (622.5)
Statistical Analysis 1: Comparison: Premarin vs Placebo; Test type: Superiority or Other; p = 0.22, t-test, 2 sided

4. Primary Outcome: Vaginal Wall Composition: Muscularis (Per-Protocol)
Description: Will assess vaginal wall histology - thicknesses of muscularis
Time Frame: Time of surgery, i.e. after 6-8 weeks of intervention
Population: as for outcome 2
Measure: Mean (Standard Error); unit: microns
Arm/Group | Premarin | Placebo
Number analyzed (Participants) | 8 | 12
microns | 7570.7 (3193.1) | 2807.1 (622.5)
Statistical Analysis 1: Comparison: Premarin vs Placebo; Test type: Superiority or Other; p = 0.088, t-test, 2 sided; t(18)=1.78, p=0.088

5. Primary Outcome: hCOL1A1, Per-Protocol
Description: Data represent ratio of total mRNA relative to postmenopausal external control.
Time Frame: Time of surgery, i.e. after 6-8 weeks of intervention
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Premarin | Placebo
Number analyzed (Participants) | 8 | 12
ratio | 2.19 [1.52 to 2.91] | 0.37 [0.18 to 0.70]
Statistical Analysis 1: Comparison: Premarin vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Serum Estrone Levels, Baseline
Time Frame: Baseline
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Premarin | Placebo
Number analyzed (Participants) | 15 | 15
pg/mL | 18.0 (2.3) | 18.5 (3.9)
Statistical Analysis 1: Comparison: Premarin vs Placebo; Test type: Superiority or Other; p = 0.91, t-test, 2 sided — t(28)=0.11, p=0.91

7. Primary Outcome: Total Collagen Content in Vaginal Muscularis, (Per-Protocol)
Description: Will assess hydroxy-proline assays as index of amount of collagen
Time Frame: Time of surgery, i.e. after 6-8 weeks of intervention
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg collagen per mg muscularis wet weight
Arm/Group | Premarin | Placebo
Number analyzed (Participants) | 8 | 12
mg collagen per mg muscularis wet weight | 302.6 (146.1) | 94.86 (29.86)
Statistical Analysis 1: Comparison: Premarin vs Placebo; Test type: Superiority or Other; p = 0.10, t-test, 2 sided — t(18)=1.69, p=.10

8. Primary Outcome: Vaginal Wall Degradative Activity, Muscularis, MMP-9
Description: Will assess zymograms for total matrix metalloprotease (MMP) 9 activity
Time Frame: Time of surgery, i.e. after 6-8 weeks of intervention
Population: All specimens with sufficient amount of tissue available for zymography analysis were used.
Measure: Mean (Standard Error); unit: Relative Units/mg protein
Arm/Group | Premarin | Placebo
Number analyzed (Participants) | 7 | 8
Relative Units/mg protein | 37.03 (15.06) | 132.34 (35.48)
Statistical Analysis 1: Comparison: Premarin vs Placebo; Test type: Superiority or Other; p = 0.020, t-test, 2 sided — t(10)=2.76, p=0.020

9. Secondary Outcome: Serum Estrone Levels, Surgery
Time Frame: Time of surgery
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Premarin | Placebo
Number analyzed (Participants) | 12 | 13
pg/mL | 22.8 (3.5) | 24.9 (6.5)
Statistical Analysis 1: Comparison: Premarin vs Placebo; Test type: Superiority or Other; p = 0.78, t-test, 2 sided — t(23)=0.28, p=0.78

10. Secondary Outcome: Serum Estradiol Levels, Baseline
Time Frame: Baseline
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Premarin | Placebo
Number analyzed (Participants) | 15 | 15
pg/mL | 11.1 (3.7) | 8.4 (1.6)
Statistical Analysis 1: Comparison: Premarin vs Placebo; Test type: Superiority or Other; p = 0.51, t-test, 2 sided — t(28)=0.67, p=0.51

11. Secondary Outcome: Serum Estradiol Levels, Surgery
Time Frame: Time of surgery
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Premarin | Placebo
Number analyzed (Participants) | 12 | 13
pg/mL | 7.8 (1.3) | 11.6 (2.7)
Statistical Analysis 1: Comparison: Premarin vs Placebo; Test type: Superiority or Other; p = 0.24, t-test, 2 sided — t(23)=1.23, p=0.24

12. Primary Outcome: Vaginal Wall Composition: Lamina Propria (Intention to Treat)
Description: Will assess vaginal wall histology - thickness of lamina propria.
Time Frame: Time of surgery, i.e. after 6-8 weeks of intervention
Measure: Mean (Standard Error); unit: microns
Arm/Group | Premarin | Placebo
Number analyzed (Participants) | 12 | 12
microns | 1042.3 (169.8) | 895.1 (153.3)
Statistical Analysis 1: Comparison: Premarin vs Placebo; Test type: Superiority or Other; p = 0.53, t-test, 2 sided

13. Primary Outcome: Vaginal Wall Composition: Lamina Propria (Per-Protocol)
Description: Will assess vaginal wall histology - thickness of lamina propria
Time Frame: Time of surgery, i.e. 6-8 weeks of intervention
Measure: Mean (Standard Error); unit: microns
Arm/Group | Premarin | Placebo
Number analyzed (Participants) | 8 | 12
microns | 1133.4 (166.2) | 895.1 (153.3)
Statistical Analysis 1: Comparison: Premarin vs Placebo; Test type: Superiority or Other; p = 0.33, t-test, 2 sided

14. Primary Outcome: hCOL3, (Per-Protocol)
Description: Data represent ratio of total mRNA relative to postmenopausal external control.
Time Frame: Time of surgery, i.e. after 6-8 weeks of intervention
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Premarin | Placebo
Number analyzed (Participants) | 8 | 12
ratio | .92 [.6 to 1.44] | .37 [.18 to .95]
Statistical Analysis 1: Comparison: Premarin vs Placebo; Test type: Superiority or Other; p = 0.05, Wilcoxon (Mann-Whitney)

15. Primary Outcome: Lysyl Oxidase (LOX) (Per-Protocol)
Description: Data represent ratio of total mRNA relative to postmenopausal external control.
Time Frame: Time of surgery, i.e. after 6-8 weeks of intervention
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Premarin | Placebo
Number analyzed (Participants) | 8 | 12
ratio | .74 (.14) | .51 (.09)
Statistical Analysis 1: Comparison: Premarin vs Placebo; Test type: Superiority or Other; p = 0.15, t-test, 2 sided

16. Primary Outcome: LOXL1 (Per-Protocol)
Description: Data represent ratio of total mRNA relative to postmenopausal external control.
Time Frame: Time of surgery, i.e. after 6-8 weeks of intervention
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Premarin | Placebo
Number analyzed (Participants) | 8 | 12
ratio | .64 (.12) | .69 (.14)
Statistical Analysis 1: Comparison: Premarin vs Placebo; Test type: Superiority or Other; p = 0.82, t-test, 2 sided

17. Primary Outcome: Tropoelastin (Per-Protocol)
Description: Data represent ratio of total mRNA relative to postmenopausal external control.
Time Frame: Time of surgery, i.e. after 6-8 weeks of intervention
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Premarin | Placebo
Number analyzed (Participants) | 8 | 12
ratio | .78 (.24) | .69 (.11)
Statistical Analysis 1: Comparison: Premarin vs Placebo; Test type: Superiority or Other; p = 0.70, t-test, 2 sided

18. Primary Outcome: TGFB1 (Per-Protocol)
Description: Data represent ratio of total mRNA relative to postmenopausal external control.
Time Frame: Time of surgery, i.e. after 6-8 weeks of intervention
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Premarin | Placebo
Number analyzed (Participants) | 8 | 12
ratio | .61 (.13) | .81 (.11)
Statistical Analysis 1: Comparison: Premarin vs Placebo; Test type: Superiority or Other; p = 0.25, t-test, 2 sided

19. Primary Outcome: Vaginal Wall Degradative Activity, Mucosa, MMP-9
Description: Will assess zymograms for total matrix metalloprotease (MMP) 9 activity
Time Frame: Time of surgery, i.e. after 6-8 weeks of intervention
Population: All specimens with sufficient amount of tissue available for zymography analysis were used.
Measure: Mean (Standard Error); unit: Relative Units/mg protein
Arm/Group | Premarin | Placebo
Number analyzed (Participants) | 7 | 8
Relative Units/mg protein | 8.97 (1.77) | 56.73 (23.20)
Statistical Analysis 1: Comparison: Premarin vs Placebo; Test type: Superiority or Other; p = 0.06, t-test, 2 sided

20. Secondary Outcome: Estimated Blood Loss
Description: Intraoperative estimated blood loss
Time Frame: Time of surgery, i.e. after 6-8 weeks of intervention
Population: In both study arms, 13 participants did undergo surgery and, therefore, had an estimated blood loss value available for analysis. However, one patient each from both study arms did not have biopsies taken (technical considerations/ intraoperative decision or conversion from total to supracervical hysterectomy without ability to collect biopsy).
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Premarin | Placebo
Number analyzed (Participants) | 13 | 13
mL | 285 (134) | 285 (270)
Statistical Analysis 1: Comparison: Premarin vs Placebo; Test type: Superiority or Other; p = 1, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 - 8 weeks of preoperative use of vaginal estrogen (vs placebo) cream
Arm/Group | Premarin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 3/15 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Premarin (N=15) | Placebo (N=15)
Vulvovaginal pain (Reproductive system and breast disorders) | 2 (2) | 0
Annoyance with cream use (Reproductive system and breast disorders) | 1 (1) | 0

LIMITATIONS AND CAVEATS:
4 patients nonadherent to study protocol in the Premarin arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No